CLINICAL TRIAL: NCT05636618
Title: A Phase I/IIa First-in-Human Study of [212Pb]VMT-α-NET Targeted Alpha-Particle Therapy for Advanced SSTR2 Positive Neuroendocrine Tumors
Brief Title: Targeted Alpha-Particle Therapy for Advanced Somatostatin Receptor Type 2 (SSTR2) Positive Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Perspective Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VMT-α-NET-T101
Record Dates: First submitted 2022-11-15; First posted 2022-12-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Tumors Unresectable; Neuroendocrine Tumor Metastatic; Gastroenteropancreatic Neuroendocrine Tumor; Bronchial Neuroendocrine Tumor; Paraganglioma; Pheochromocytoma
Keywords: Radiopharmaceuticals; Somatostatin Receptor Type 2 (SSTR2); Neuroendocrine Tumors; Metastatic Neuroendocrine Tumors; Pb-212; Theranostics; Alpha Particle Therapy; Radiotherapy; [212Pb]VMT-α-NET; VMT-α-NET-T01; Pb-203
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Paraganglioma; Pheochromocytoma; Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: A Phase I/IIa First-in-Human Study of [212Pb]VMT-α-NET Targeted Alpha-Particle Therapy for Advanced SSTR2 Positive Neuroendocrine Tumors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Finding (Experimental): Dose Finding to determine OBD and potential RP2D in up to 200 patients receiving up to 4 administrations of [212Pb]VMT-α-NET approximately 8 weeks apart.
  A dosimetry sub-study utilizing [203Pb]VMT-α-NET is incorporated into the study.
  Interventions: Drug: [203Pb]VMT-α-NET; Drug: [212Pb]VMT-α-NET
- Dose Expansion (Experimental): Dose with up to 60 subjects at RP2D for further assessment of safety and preliminary efficacy.
  Interventions: Drug: [203Pb]VMT-α-NET; Drug: [212Pb]VMT-α-NET

INTERVENTIONS:
Drug: [203Pb]VMT-α-NET — [203Pb]VMT-α-NET is administered by intravenous bolus injection for single-photon emission computed tomography imaging.
Drug: [212Pb]VMT-α-NET — [212Pb]VMT-α-NET is administered by intravenous infusion for treatment of SSTR2 expressing neuroendocrine tumors.

SUMMARY:
This study is Phase I/IIa First-in-Human Study of [212Pb]VMT-α-NET Targeted Alpha-Particle Therapy for Advanced SSTR2 Positive Neuroendocrine Tumors

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, radioactivity dose-finding/ dose expansion study of [212Pb]VMT-α-NET in up to 260 adult subjects with unresectable or metastatic SSTR2-expressing neuroendocrine tumors (NETs) who have not received prior peptide receptor radionuclide therapy (PRRT).

Somatostatin Receptor type 2 (SSTR2) is highly expressed on various tumors including NETs and therefore is an attractive therapeutic target for NET treatment. Lead-212 ([212Pb]-) based peptide-radiopharmaceuticals are an emerging class of targeted alpha-particle cancer therapies that have potential to improve delivery of a highly effective form of radiation.

[212Pb] VMT-a-NET is a targeted alpha therapy agent designed to enhance the precision and effectiveness of cancer treatment by delivering a highly potent form of radiation directly to cancer cells. This approach aims to maximize radiation delivery to tumors while minimizing exposure to healthy tissues.

The study will be conducted in 2 parts:

Part 1: Phase I Dose-Finding: Subjects will receive radioactive doses of [212Pb]VMT-α-NET up to a maximum dose of 222 MBq (6 mCi) for dose-limiting toxicity (DLT) observation, determining Optimal Biological Dose (OBD) and potential Recommended Phase 2 Dose (RP2D) for Part 2 (Dose Expansion). Dose changes or adjustments will be made by the safety monitoring committee (SMC) and Sponsor.

The RP2D will be determined following a holistic analysis of observed DLTs, adverse events (AEs), estimated cumulative organ radiation exposure, and efficacy signals over the course of all treatment cycles for all dose cohorts.

Part 2: Phase IIa Dose-Expansion: This part will enroll subjects who will receive RP2D identified in Part 1 for further assessment of safety and preliminary efficacy.

Reno-protective amino acids will be co-administered prior to each [212Pb]VMT-α-NET dose in all subjects. Dose-finding will be based on an adaptive design until optimal biologic dose is identified or the pre-specified rules are met.

A dosimetry sub-study using [203Pb]VMT-α-NET will be conducted. The subjects will undergo dosimetric evaluation prior to receiving the therapeutic agent.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (ages ≥18) PRRT-naïve subjects with NETs by local pathology.
2. Locally advanced/unresectable or metastatic NETs.
3. Radiological evidence of measurable disease by RECIST v1.1 criteria on CT with contrast or MRI of the areas of tumor involvement within 60 days of enrollment.
4. Lesions must have shown radiological evidence of disease progression in the 12 months prior to enrollment.
5. Demonstration of lesional SSTR2 expression using an FDA-approved somatostatin receptor PET imaging agent, e.g. [68Ga]DOTATATE, [64Cu]DOTATATE, or [68Ga]DOTATOC, (SSTR2 positivity defined as uptake > background liver) obtained and interpreted in accordance with product labeling and appropriate clinical use criteria within 12 months of enrollment.
6. ECOG Performance Status ≤ 1.
7. Subjects with HIV positivity are allowed if CD4 Count > 350 cells/μL.
8. Concurrent Somatostatin Analog (SSA) Therapy use while on protocol therapy is allowed provided that the subject the subject must be able to tolerate withholding long-acting SSA therapy for a minimum of 28 days and short-acting SSA therapy for a minimum of 24 hours before the first and subsequent administrations of [203Pb]VMT-α-NET or [212Pb]VMT-α-NET
9. Progressive Disease on approved therapies other than radionuclide therapy.
10. Must have clinically demonstrated adequate catecholamine blockade if catecholamine-secreting pheochromocytoma/paraganglioma tumors are present.
11. Able to understand and sign informed consent and comply with all study requirements.
12. Life expectancy > 3 months.
13. Satisfactory organ function as determined by laboratory testing.
14. For females of reproductive potential: agree to use of highly effective contraception and refrain from donating eggs (ova, oocytes) for the purpose of reproduction starting from screening, during treatment, and for at least 6 months after the last dose of [212Pb]VMT-α-NET
15. For males of reproductive potential: agree to use of condoms or other methods to ensure effective contraception with partner and refrain from donating sperm starting from screening, during treatment, and for at least 6 months after the last dose of [212Pb]VMT-α-NET

Exclusion Criteria:

1. Known hypersensitivity to SSA, SSTR imaging agents or any of the excipients of [212Pb]VMT-α-NET.
2. Active secondary malignancy.
3. Pregnancy or breastfeeding a child.
4. Febrile illness within 48 hours of any scheduled [212Pb]VMT-α-NET administration should be rescheduled > 48 hours after resolution of fever].
5. Treatment with another investigational medicinal product within 30 days of anticipated treatment.
6. Prior treatment with systemic PRRT based therapies (i.e., [90Y] DOTATATE/DOTATOC or [177Lu] DOTATATE)
7. Prior treatment with 90-Yttrium radioembolization must be completed at least 6 months prior to enrollment.
8. External beam radiation therapy must be completed at least 30 days prior to enrollment.
9. Prior treatment with systemic anticancer therapy must be completed at least 30 days prior to enrollment (except for SSAs in subjects with functional tumors).
10. Major surgery must be completed at least 30 days prior to enrollment.
11. Known brain metastases; unless these metastases have been treated and stabilized 6 months prior to enrollment and the subject has been off steroid support for at least 14 days prior to enrollment.
12. Recently diagnosed and active infections requiring a time-limited course of antifungals or antibiotics in the 3 days prior to enrollment.
13. Receipt of live attenuated vaccines in the 7 days prior to enrollment.
14. Grade 3 nausea/vomiting or diarrhea within 72 hours before the of first scheduled dose of [212Pb]VMT-α-NET despite adequate antiemetic and other supportive care
15. Known medical condition which would make this protocol unreasonably hazardous for the subject.
16. Medical history of a condition resulting in a severe allergic reaction such as anaphylaxis or angioedema to known components of the Investigational Medicinal Product or excipients.
17. Current abuse of alcohol or illicit drugs (exclusive of use of medically prescribed cannabinoids).
18. Existence of any medical or social issues likely to interfere with study conduct or that may cause increased risk to the subject or to others, e.g., lack of ability to follow radiation safety precautions.
19. QTc > 450 milliseconds for males and females.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2029-11-26 (Estimated); Study Completion 2029-12-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) after the first administration of [212Pb]VMT-α-NET | Incidence and severity of DLTs during the first 42 days of study treatment will be assessed.
  DLTs describe side effects of a drug that are serious enough to prevent an increase in dose
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 | Up to week 96
  Percentage of subjects with complete responses (CRs) or partial responses (PRs) to at least 1 administration of [212Pb]VMT-α-NET
Number of subjects with adverse events (AEs) | Until the end of study (3 years after end-of-study visit)
  Any untoward medical occurrence in a clinical investigational participant administered [212Pb]VMT-α-NET and which does not necessarily have a causal relationship with this treatment. Associated Adverse Events (AE) or Serious AEs are assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Anti-tumor efficacy of [212Pb]VMT-α-NET in terms of tumor response | Until the end of study (3 years after end-of-study visit)
  Determination of the overall response rate (ORR) by RECIST v1.1 in subjects with neuroendocrine tumors
Determine the duration of response (DOR) receiving [212Pb]VMT-α-NET. | Up to week 96
  The length of time that a tumor continues to respond to treatment without the cancer growing or spreading determined by RECIST v1.1
Determination of Progression-free survival (PFS) | Up to week 96
  PFS is how long a subject lives without the disease worsening as evaluated by RECIST v1.1
To investigate the Overall Survival (OS) following treatment with [212Pb]VMT-α-NET | Until the end of study (3 years after end-of-study visit)
  OS is how long a subject lives after a subject starts treatment
Determination of pharmacokinetic properties of [212Pb]VMT-α-NET. | 24 hours following [212Pb]VMT-α-NET dosing.
  Blood radioactivity pharmacokinetic parameter i.e. area under the plasma concentration versus time curve (AUC) is determined.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Mayo Clinic, Jacksonville, Florida
  - Biogenix Molecular, Miami, Florida
  - The University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - BAMF Health, Grand Rapids, Michigan
  - Michigan Health Professionals, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Protocol, CSR